CLINICAL TRIAL: NCT01556932
Title: A Randomized Trial of the Effectiveness of Topical "ABH Gel" (Ativan®, Lorazepam; Benadryl®, Diphenhydramine; and Haldol®, Haloperidol Gel) Versus Placebo in Patients With Nausea
Brief Title: Randomized Trial of the Effectiveness of Topical "ABH Gel" vs. Placebo in Cancer Patients With Nausea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: MCC-14141; NCI-2012-00220 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-03-13; First posted 2012-03-19 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Lorazepam; Diphenhydramine; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo then ABH (Experimental): All subjects randomized to two sequences of treatments: either placebo-ABH or ABH-placebo. All participants will receive both drug A and drug B.
  After applying gel, Drug A or B, on wrists for 2 minutes, time 0. From baseline to 60 minutes of treatment two options will occur. At 60 minutes, if patients have at least 1 point reduction in their nausea score, they must wait 4 hours before switching to opposite drug. After administration of drug, the study procedures will be repeated. Or, at 60 minutes, if no change or increase in nausea score has been recorded, alternative treatment will be given. If the second treatment is ineffective at one hour (total time 2 hours) then alternative usual medications will be given. After completion of study treatment, patients are followed up for up to 8 hours.
  Interventions: Drug: ABH gel; Other: placebo
- ABH then placebo (Experimental): All subjects randomized to two sequences of treatments: either placebo-ABH or ABH-placebo. All participants will receive both drug A and drug B.
  After applying gel, Drug A or B, on wrists for 2 minutes, time 0. From baseline to 60 minutes of treatment two options will occur. At 60 minutes, if patients have at least 1 point reduction in their nausea score, they must wait 4 hours before switching to opposite drug. After administration of drug, the study procedures will be repeated. Or, at 60 minutes, if no change or increase in nausea score has been recorded, alternative treatment will be given. If the second treatment is ineffective at one hour (total time 2 hours) then alternative usual medications will be given. After completion of study treatment, patients are followed up for up to 8 hours.
  Interventions: Drug: ABH gel; Other: placebo

INTERVENTIONS:
Drug: ABH gel — Given topically
  Other Names: Ativan; lorazepam; diphenhydramine hydrochloride; Benadryl; Bendylate; Eldadryl; SK-Diphenhydramine; haloperidol; Haldol; McN-JR-1625; R-1625
Other: placebo — Given topically
  Other Names: PLCB

SUMMARY:
This randomized clinical trial studies ABH (lorazepam, diphenhydramine hydrochloride, and haloperidol) gel in patients with nausea. ABH gel, when absorbed into the skin, may be an effective treatment for nausea and vomiting. The general purpose of this research study is to improve the treatment of nausea and vomiting.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary outcome is the change in numeric rating scale in self-reported nausea on a 0-10 scale from baseline to 60 minutes of treatment.

OUTLINE: All individuals who are eligible are randomized to a sequence of treatments: either placebo-ABH or ABH-placebo. The randomization list will be generated by the Study Biostatistician. Neither the patient nor the investigator will have knowledge of the actual content of Drug A or B, so the study will be double-blinded, and placebo controlled.

Drug A: The dose of the drugs in the 1.0 mL dose will be 2 mg of lorazepam, 25 mg of diphenhydramine, and 2 mg of haloperidol in a pluronic lecithin organogel. It will be rubbed on the volar surface of the wrists by the subject, for 2 minutes as done in clinical practice, at time 0. Drug B: equivalent but no ABH.

Subjects will rub 1 mL of the first drug, Drug A gel, between their wrists for 2 minutes.

Subjects will be asked to rate and complete their nausea on the Memorial Symptom Assessment Scale (CMSAS). At time 60 two options can occur. One, if there is no effect after the first drug in one hour, then patients will receive the second drug. If there is no effect in one hour from second drug, patients will stop the study and resume normal treatment for their nausea. Or two, if the first gel reduces nausea by more than 1 point on the 0-10 scale, subjects will wait 4 hours to apply the next gel. At this point, the study procedures will be repeated. After treatment, patients are followed up for up to 8 hours.

Subjects will be asked to rate their nausea on a 0 (no nausea) to 10 (worst possible nausea) scale at baseline, 60, 120, 180, and 240 minutes.

Subjects will complete the Memorial Symptom Assessment Scale (CMSAS), a reliable and valid instrument for assessing relevant symptoms including lack of energy, lack of appetite, pain, dry mouth, weight loss, feeling drowsy, shortness of breath, constipation, difficulty sleeping, difficulty concentrating, and nausea.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* No allergies to the drugs
* Able to complete the forms
* If a woman of childbearing age, agree to use contraception; women will be offered a pregnancy test before doing the trial if they request one, as stated in the Informed Consent Form
* Patients must have a self reported nausea score of at least 4 on a numeric rating scale of 0-10 (zero being no nausea and ten being the worst possible nausea); patients are not required to have vomiting
* Patients must have had or have cancer, or have had a consultation with the palliative care team
* They must not have had any changes to their nausea program within the past 12 hours, if on anti-emetics
* Patients must not have received chemotherapy within 5 days, unless it is a stable oral chemotherapy drug such as capecitabine (Xeloda), erlotinib (Tarceva), or similar

Exclusion Criteria:

* History of substance abuse, psychiatric disorder, acquired brain injury, the possibility of pregnancy (not using birth control, and of child bearing age)
* Use of any medication that would contraindicate benzodiazepine administration
* Pregnant or nursing
* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devon Fletcher, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from Massey Cancer Center, in Richmond City, Virginia USA between March 2012 until May 2013.
Pre-assignment Details: 25 participants were consented to the research study. Two of them no longer were nauseous and never started treatment. One subject expired on the study. 22 subjects enrolled but only 20 evaluable subjects' data was completed for analysis.
Groups:
- ABH Gel- Placebo: All individuals who are eligible were randomized to a sequence of treatments: either placebo-ABH or ABH-placebo. All participants were on one arm but separate sequences because they started on different drugs. This group started with ABH gel first and then went to Placebo.The randomization list will be generated by the Study Biostatistician.
- Placebo-ABH Gel: All individuals who are eligible were randomized to a sequence of treatments: either placebo-ABH or ABH-placebo. All participants were on one arm but separate sequences because they started on different drugs. This group started with Placebo first and then went to ABH gel. The randomization list will be generated by the Study Biostatistician.
Period: Baseline First Treatment
Arm/Group | ABH Gel- Placebo | Placebo-ABH Gel
Started | 13 | 9
Recieved | 13 | 9
Completed | 13 | 9
Not Completed | 0 | 0
Period: Time Point 60 Minutes
Arm/Group | ABH Gel- Placebo | Placebo-ABH Gel
Started | 13 (1 subject withdrew and never started second treatment.) | 9 (1 subject withdrew and never started second treatment.)
Recieved | 12 | 8
Completed | 12 | 8
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Treament
Arm/Group | ABH Gel- Placebo | Placebo-ABH Gel
Started | 12 | 8
Recieved | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients who were eligible were randomly assigned to two sequences: one group used ABH gel first and then the placebo; and the other group used the placebo first and then ABH gel. We assumed there was no carry-over effect from the first treatment to the second. In total, 22 patients were enrolled but 20 subjects completed the study.
Groups:
- All Participants: All participants go through Placebo-ABH or ABH-placebo depending on the sequence they were randomized to. Patients are randomized into Placebo-ABH or ABH-Placebo sequence.
  Sequence 1:Patients apply Drug A gel topically for 2 minutes at time 0. After 1 hour, if no change or increase in the nausea score alternative treatment will be given Drug B. If the second treatment is ineffective at one hour (total time 2 hours) alternative usual medications will be given Drug A. ABH is Ativan (lorazepam), Benadryl (diphenhydramine), and Haldol.
  Sequence 2:Patients will apply Drug B gel topically for 2 minutes at time 0. After 1 hour, if no change or increase in the nausea score alternative treatment will be given Drug A. If the second treatment is ineffective at one hour (total time 2 hours) alternative usual medications will be given Drug B. ABH is Ativan (lorazepam), Benadryl (diphenhydramine), and Haldol.
Arm/Group | All Participants
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1600 (14.1500294)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: The Change in Numeric Rating Scale in Self-reported Nausea From Baseline Minus 60 Minutes of Treatment.
Description: The outcome measure for change was calculated from value at baseline minus value at 60 minutes. Subjects were asked to rate their nausea on a 0 (no nausea) to 10 (worst possible nausea) scale. Subjects who were eligible were randomly assigned to two sequences: one sequence used ABH gel first and then placebo; and the other sequence used placebo first and then ABH gel. We assumed that there was no carry-over effect from the first treatment to the second. A paired t-test was used to compare if ABH gel is not better than the placebo gel. A repeated measure analysis was used to compare the two treatment sequences. This endpoint was chosen as the drug gel because it is typically used as a "prn" (as needed) gel in actual practice, when relief is needed in short order.
Time Frame: 60 minutes after application
Population: 25 participants were consented, two subjects declined treatment, one expired subject. Two subjects refused to continue after first treatment and did not complete the second treatment. Only 20 patients were analyzed because of missing data not done by those two subjects on the second treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ABH Gel: ABH Gel applied topically for 2 minutes.
- Placebo: Placebo applied topically for 2 minutes.
Arm/Group | ABH Gel | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | 1.70 (2.05) | 0.90 (2.47)
Statistical Analysis 1: Comparison: ABH Gel vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.8, Standard Deviation 3.2541

ADVERSE EVENTS:
Time Frame: Adverse event data was measured at 5 time points for each patient. Following times: prior (time 0), 60, 120, 180, and 240 minutes after the gel. Total AE reporting was 1 year and 3 months.
Groups:
- Arm A and Arm B: Patients apply lorazepam, diphenhydramine hydrochloride, and haloperidol gel topically over 2 minutes and placebo topically over 2 minutes.
Arm/Group | Arm A and Arm B
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes